CLINICAL TRIAL: NCT04328740
Title: A Phase I, First-in-human, Open-label, Dose Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Oral TP 1454
Brief Title: Phase 1 Study of Oral TP-1454
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TP-1454-101
Record Dates: First submitted 2020-03-20; First posted 2020-03-31 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor; Anal Cancer
Keywords: Sumitomo Pharma Oncology; Phase 1; Advanced Solid Tumors; Refractory; Anal cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TP-1454 (Experimental): Flat dose once or twice daily
  Interventions: Drug: TP-1454 monotherapy

INTERVENTIONS:
Drug: TP-1454 monotherapy — Flat dose once or twice daily, alone

SUMMARY:
This study will evaluate the safety and tolerability of oral TP-1454 in patients with advanced metastatic or progressive solid tumors and anal cancer.

DETAILED DESCRIPTION:
Primary Objective:

• To establish the MTD and/or Recommended Phase 2 Dose (RP2D) of orally administered TP-1454 in patients with metastatic solid tumors and anal cancer.

Secondary Objectives:

* To establish the pharmacokinetic (PK) profile of orally administered TP-1454
* To observe patients for any evidence of antitumor activity of TP 1454 by objective radiographic assessment
* To assess the safety and tolerability of TP-1454

ELIGIBILITY:
Inclusion Criteria:

1. Patients to be enrolled during Dose Escalation with capsules must have a histologically confirmed diagnosis of advanced metastatic or progressive solid tumor who are refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition (enrollment complete).
2. Following approval of Amendment 5.0, patients to be enrolled during Dose Escalation with Tablets must have a histologically confirmed diagnosis of anal cancer and:

   1. have received at least one line of systemic platinum-based therapy in the advanced setting; (Note: Systemic platinum therapy given in the adjuvant setting will meet this criterion if there is recurrence or metastasis within 6 months of completing adjuvant therapy.); and
   2. have received no more than 3 total lines of systemic therapy in the advanced setting.
3. Have measurable disease as outlined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
5. Be ≥18 years of age
6. Have a negative pregnancy test (if female of childbearing potential)
7. Have acceptable liver function:

   1. Bilirubin ≤1.5x upper limit of normal (ULN) (unless associated with Gilbert syndrome)
   2. Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) and alkaline phosphatase ≤2.5x ULN* *If liver metastases are present, then ≤ 3x ULN is allowed.
8. Have acceptable renal function: calculated creatinine clearance ≥60 mL/min (using Cockcroft Gault formula)
9. Have acceptable hematologic status:

   1. Granulocyte ≥1500 cells/mm3
   2. Platelet count ≥100,000 (plt/mm3)
   3. Hemoglobin ≥8 g/dL
10. Have acceptable coagulation status:

    1. International Normalized Ratio (INR) or Prothrombin time (PT) within 1.5x normal limits unless the patient is receiving anticoagulant therapy, in which case, the patient's PT or partial thromboplastin time (PTT) must be within the therapeutic range of intended use for their anticoagulant.
    2. Partial activated partial thromboplastin time (aPTT) or activated partial thromboplastin time (aPTT) within 1.5x normal limits unless the patient is receiving anticoagulant therapy, in which case, the patient's PT or PTT must be within the therapeutic range of intended use for their anticoagulant.
11. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use a highly effective method of contraception prior to study entry for the duration of study participation and for at least 3 months (males) and 6 months (females) after the last study drug dose.
12. Male patients only: must agree not to donate sperm during the study and for 3 months after the last dose of TP-1454.
13. Women of childbearing potential must agree not to donate eggs during the study and for 6 months after the last dose of TP-1454.
14. Have read and signed the Institutional Review Board (IRB)-approved informed consent form (ICF) prior to any study-related procedure. (In the event that the patient is rescreened for study participation or a protocol amendment alters the care of an ongoing patient, a new ICF must be signed.)
15. Dose escalation in mSCCA with tablets only: Patients who are HIV+ may be enrolled if the following conditions are met:

    1. CD4+ T-cell count ≥ 300/µL
    2. No opportunistic infection within the past 12 months
    3. Treatment with established antiretroviral therapy for at least 4 weeks with a viral load < 400 copies/mL prior to first dose with TP-1454.
16. Dose escalation in mSCCA with tablets only: Patients who have had hepatitis B or C viral infections (HBV or HCV, respectively) may be enrolled if the following conditions are met:

    1. Have completed or are undergoing curative antiviral treatment with viral load below the limit of quantification
    2. Test positive for antibody and negative for viral RNA

Exclusion Criteria:

1. New York Heart Association Class III or IV cardiac disease, or myocardial infarction, severe unstable angina, coronary/peripheral artery bypass graft, congestive heart failure within the past 6 months or evidence of ischemia on electrocardiogram (ECG) within 14 days prior to Cycle 1/Day 1
2. Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of >450 msec in men and >470 msec in women
3. Have a seizure disorder requiring anticonvulsant therapy
4. Have untreated central nervous system (CNS) metastases including carcinomatous meningitis. Patients with definitively treated (radiotherapy or surgery) CNS metastases may be eligible if asymptomatic and not receiving corticosteroids in excess of prednisone 10 mg (or equivalent) per day for ≥2 weeks before first dose of TP-1454
5. Have hypoxemia (defined as resting O2 saturation of ≤90% breathing room air)
6. Have symptomatic interstitial lung disease
7. Have undergone major surgery within 2 weeks prior to Cycle 1/Day 1
8. Have active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
9. Are pregnant or nursing
10. Received treatment with radiation therapy to a target lesion, surgery, chemotherapy, or investigational therapy within 28 days or 5 half-lives, whichever occurs first, prior to study entry (6 weeks for nitrosoureas or mitomycin C)
11. Are unwilling or unable to comply with procedures required in this protocol
12. Dose escalation in solid tumors with capsules only: Have known infection with hepatitis B, or hepatitis C. Patients with history of chronic hepatitis that is currently not active are eligible
13. Have a serious nonmalignant disease (eg, hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor
14. Are currently receiving any other investigational agent
15. Have exhibited allergic reactions to a similar structural compound, biological agent, or formulation(s)
16. Have malabsorption conditions or have undergone significant surgery to the gastrointestinal tract that could impair absorption or that could result in short bowel syndrome with diarrhea due to malabsorption
17. Have a history of malignancy within the past 24 months except curatively treated in situ cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) | 50 months
  MTD will be determined based upon toxicity grades which are defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 5.0.
Determine recommended Ph2 dose (RP2D) of TP-1454 | 50 months
  To establish the RP2D for future studies with TP-1454. MTD, PK and PD data to be reviewed.
Incidence of SAEs and AEs resulting in study discontinuation, as assessed by NCI NTCAE v5.0 | From date of treatment through 30 days after End of Treatment, an average of 6 months
  With approval of protocol amendment 7, the primary objective of this study is to continue to monitor the safety and tolerability of TP-1454 in ongoing patients.

SECONDARY OUTCOMES:
Determine incidence of dose-limiting toxicities (DLTs) | 28 days
  A DLT is defined as a drug-related toxicity that is observed to occur within the first 28 days
Determine antitumor activity of TP-1454. | 50 months
  Objective radiographic assessment to be performed to determine antitumor activity by Response Evaluation Criteria in Solid Tumors (RECIST criteria v 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (11):
- United States (11):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Southern California - Norris Cancer Center and Hoag Memorial Hospital, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Vanderbilt University, Nashville, Tennessee
  - Texas Oncology Baylor Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No